CLINICAL TRIAL: NCT04450511
Title: Combined Effect of Pelvic Floor Magnetic Stimulation and Bladder Training in Women With Idiopathic Overactive Bladder: A Prospective Randomised Controlled Trial
Brief Title: Pelvic Floor Magnetic Stimulation in Women With Idiopathic Overactive Bladder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Necmettin Yildiz, Professor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 60116787-020/37878
Record Dates: First submitted 2020-06-25; First posted 2020-06-29 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Urge Incontinence Episodes After the Magnetic Stimulation Added to Bladder Training in Women With Idiopathic Overactive Bladder
Keywords: idiopathic overactive bladder; bladder training; magnetic stimulation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Bladder Training (BT) (Active Comparator): BT, consisting of four stages, did not contain any PFM training programs in all groups. In these stages, including urgency suppression strategies, it was aimed to delay urination, to inhibit detrusor contraction and to prevent urgency; by squeezing the PFM several times in a row (women were encouraged to pause/stop their work, sit down if possible, relax the entire body and squeeze PFM repeatedly), breathing deeply, giving their attention to another job for a while and self-motivating (I can do it, I can check the urination, etc.).
  Interventions: Other: Bladder Training (BT)
- Group 2: Bladder Training+Magnetic Stimulation (Experimental): Patients are told to sit on the chair with a magnetic coil below the chair. When a volume conductor is inserted by this magnetic ﬁeld, an eddy current ﬂow is generated. This eddy current stimulates nerve or muscle of the pelvic ﬂoor. To apply MS, the device was set to generate its maximum stimuli, with a stimulation pulse width of 200 μs and a stimulation repetition cycle of 10 Hz in accordance with the literature. When setting the device at each treatment session, patients were interviewed so that they received stimuli at the maximum stimulation intensity (maximum tolerable stimulation intensity) .
  Interventions: Device: Magnetic stimulation -Armchair type (MS); Other: Bladder Training (BT)

INTERVENTIONS:
Device: Magnetic stimulation -Armchair type (MS) — MS was applied two days a week, 20 minutes a day, a total of 12 sessions for 6 weeks.
  Other Names: Extracorporeal magnetic stimulation
  Arms: Group 2: Bladder Training+Magnetic Stimulation
Other: Bladder Training (BT) — Bladder Training (BT)

SUMMARY:
In clinical practice, Bladder Training (BT) and Magnetic stimulation (MS) are frequently used together in the treatment of women with idiopathic overactive bladder (OAB). Up to our knowledge, there is no study evaluating the combined effect of magnetic stimulation and bladder training in women with idiopathic OAB in the literature. Moreover, there is no recommendation on conservative treatment combinations in the guidelines due to insufficient data. At this stage, studies are needed to determine whether it will be effective to use MS in combination with other conservative treatment options. In addition, in the light of our clinical experience, we think that this issue is still open for research. In our study, adding MS to BT in women with idiopathic OAB is thought to contribute additionally to the efficacy of treatment with BT.

Our study is the first prospective randomized controlled trial that compares the efficacy of BT and BT plus MS in women with idiopathic OAB. In this study, we aimed to evaluate the efficacy of MS added to BT on incontinence-related QoL and clinical parameters in women with idiopathic OAB.

DETAILED DESCRIPTION:
This study is a prospectively randomized, controlled trial. The trial is held at Urogynecological Rehabilitation Unit of University Hospital, Physical Medicine and Rehabilitation Department between September 2020 and November 2021. The local ethics committee approve the study (approval no: 60116787-020/37878). Patients are informed about the purpose and contents of the study and all women give written consent to participate.

By using a random number generator, all patients which included the study were randomized into two groups as follows: The Group 1 received BT program alone, the Group 2 received BT plus MS.

Group 1: Bladder Training (BT) - Control group All women were informed about BT for 30 minutes. Then it was given as a written brochure to be implemented as a home program.

BT, consisting of four stages, did not contain any pelvic floor muscle (PFM) training programs in two groups.

Group 2: BT plus MS Patients are told to sit on the chair with a magnetic coil below the chair. When a volume conductor is inserted by this magnetic ﬁeld, an eddy current ﬂow is generated. This eddy current stimulates nerve or muscle of the pelvic ﬂoor. To apply MS, the device was set to generate its maximum stimuli, with a stimulation pulse width of 200 μs and a stimulation repetition cycle of 10 Hz in accordance with the literature (10,13-15). When setting the device at each treatment session, patients were interviewed so that they received stimuli at the maximum stimulation intensity (maximum tolerable stimulation intensity) (10). MS was applied two days a week, 20 minutes a day, a total of 12 sessions for 6 weeks. MS sessions were performed by other physician.

ELIGIBILITY:
Inclusion Criteria:

1. Women over the age of 18 with clinical diagnosis of idiopathic OAB
2. Urodynamically confirmed detrusor overactivity (the presence of detrusor contractions in the ﬁlling phase of saline cystometry)
3. Not tolerated or unresponsive to antimuscarinics and discontinued at least 4 weeks
4. Able to give written, informed consent
5. Able to understand the procedures, advantages and possible side effects
6. Willing and able to complete the voiding diary and QoL questionnaire
7. The strength of PFM 3/5 and more

Exclusion Criteria:

1. History of BT, MS therapy
2. Pregnancy or intention to become pregnant during the study
3. Current vulvovaginitis or urinary tract infections or malignancy
4. More than stage 2 according to the pelvic organ prolapse quantification
5. Cardiac pacemaker, implanted defibrillator, coronary artery stent
6. Ongoing treatment for arrhythmia
7. Lower abdominal pain or dysmenorrhea yet to be diagnosed
8. Electronic device or metallic implant applied to areas between the lumbar region and lower extremities
9. Previous urogynecological surgery within 3 months
10. Ongoing surgical treatment or treatment with implantable devices for urinary incontinence or use of intrauterine copper devices
11. Neurogenic bladder, signs of neurologic abnormalities at objective examination; history of the peripheral or central neurologic pathology
12. Ultrasonographic evidence of post voiding residual volume more than 100 ml

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women over the age of 18 with clinical diagnosis of idiopathic OAB and urodynamically conﬁrmed detrusor overactivity (the presence of detrusor contractions in the ﬁlling phase of saline cystometry)
Enrollment: 76 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-11-29 (Actual)

PRIMARY OUTCOMES:
Incontinence episodes | 6 weeks
  Patients with a 50% or greater reduction in incontinence episodes were consider positive responders

SECONDARY OUTCOMES:
Severity of incontinence | 6 weeks
  The 24-hour pad test was carried out to evaluate urinary loss.
Nocturia | 6 weeks
  It was used "nocturia" from data collected with a 3-day bladder diary.
Frequency | 6 weeks
  It was used "frequency" from data collected with a 3-day bladder diary.
Number of pads | 6 weeks
  It was used "number of pads" from data collected with a 3-day bladder diary.
Symptom severity | 6 weeks
  Overactive Bladder Questionnaire (OAB-V8) was used to evaluate symptom severity in patients with in the study.
QoL | 6 weeks
  The Incontinence Impact Questionnaire (IIQ-7) scale which has great validity in studies was used to assess the patient's QoL associated with incontinence problem
Sexual Functions | 6 weeks
  The Female Sexual Function Index (FSFI) is a valid, reliable, and anonymously designed ques¬tionnaire with six areas (desire, subjective arousal, lubrica¬tion, orgasm, satisfaction, pain), and includes 19 questions that measure female sexual function.
Cure and improvement rate | 6 weeks
  In 24-hour pad test, 1.3 gr under of it was considered as a cure. The improvement was assessed in terms of 50% and more reduction in wet weight compared to baseline measurements in the 24-hour pad test

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Kınıklı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No